CLINICAL TRIAL: NCT05783479
Title: Estriol and Hyaluronic Acid in Cervical Preparation for Mini-hysteroscopy in Peri- and Postmenopausal Women
Brief Title: Pharmacological Preparation of the Cervix for Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Iwona Magdalena Gawron, Ph.D., Principal Investigator, Jagiellonian University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1072.6120.128.2021
Record Dates: First submitted 2023-03-11; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Uterine Polyp; Uterine Bleeding; Endometrium; Senility
MeSH Terms: conditions — Uterine Hemorrhage | interventions — Estradiol; Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Comparison of endpoints in three study arms: i) estradiol 0.5 mg in vaginal cream twice daily for 10 days pre-procedure, ii) hyaluronic acid 5 mg in vaginal gel twice daily for 10 days pre-procedure, iii) no treatment (control).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (estradiol) (Active Comparator): estradiol 0.5 mg in vaginal cream twice daily for 10 days pre-procedure
  Interventions: Drug: estradiol
- 2 (hyaluronic acid) (Active Comparator): hyaluronic acid 5 mg in vaginal gel twice daily for 10 days pre-procedure
  Interventions: Drug: Hyaluronic acid
- 3 (control) (No Intervention): no preparation of the cervix - arm without medication

INTERVENTIONS:
Drug: estradiol — estradiol 0.5 mg in vaginal cream twice daily for 10 days pre-procedure
  Arms: 1 (estradiol)
Drug: Hyaluronic acid — hyaluronic acid 5 mg in vaginal gel twice daily for 10 days pre-procedure
  Arms: 2 (hyaluronic acid)

SUMMARY:
Pain accompanying office hysteroscopy is the most common reason for its discontinuation. Urogenital atrophy may cause technical difficulties in passage through the cervical canal, further increasing the pain. The aim was to evaluate the effectiveness of vaginal estradiol and hyaluronic acid to facilitate diagnostic hysteroscopy in peri- and postmenopausal women.

DETAILED DESCRIPTION:
A prospective cohort tertiary-center study includes women over 45 years of age subjected to office hysteroscopy in 2021-2022. Women who consent are assigned to three study arms: i) estradiol 0.5 mg in vaginal cream twice daily for 10 days pre-procedure, ii) hyaluronic acid 5 mg in vaginal gel twice daily for 10 days pre-procedure, iii) no treatment (control). The following endpoints are compared: need for cervical dilation, incidence of severe urogenital atrophy and vaso-vagal reaction, time of cervical passage, cervical canal diameter, pain during and after the procedure in the Numeric Rating Scale (NRS).

ELIGIBILITY:
Inclusion Criteria:

* age 45-90 years
* uterine cavity focal lesion, abnormal uterine bleeding

Exclusion Criteria:

* drug allergy
* no consent to the procedure or participation in the study

Ages: 45 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Intensification of pain during and after the procedure | up to 6 months
  Intensity of pain in Numeric Rating Scale (NRS: 0-10)
The need of cervical dilation | up to 6 months
  The need for cervical dilation (yes/no) to penetrate the cervix and enter the uterine cavity

SECONDARY OUTCOMES:
Cervical passage time | up to 6 months
  Cervical penetration time (minutes) from visualization of the external cervical os to reaching the uterine cavity
Occurrence of a vasovagal reaction | up to 6 months
  the occurrence of a vasovagal reaction (fall in blood pressure, bradycardia, syncope)
Occurrence of severe urogenital atrophy (paleness and thinning of the vaginal epithelium, petechiae and shallow ulcers, bleeding and contact) | up to 6 months
  Clinical evaluation of the occurrence of symptoms of urogenital atrophy

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jach, Prof., Study Chair — Jagiellonian University
Locations (1):
- Jagiellonian University Medical College, Department of Gynecology and Obstetrics, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No